CLINICAL TRIAL: NCT03694249
Title: A Pilot Trial of Ifetroban, A Thromboxane A2 Receptor Antagonist, in Patients With Malignant Solid Tumors at High Risk of Metastatic Recurrence
Brief Title: Ifetroban in Treating Patients With Malignant Solid Tumors at High Risk of Metastatic Recurrence
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sonya Reid, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VICC MD1854; NCI-2018-01930 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2018-09-24; First posted 2018-10-03 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (ifetroban) (Experimental): ifetroban capsule (250mg) will be taken by mouth daily.
  Interventions: Drug: Ifetroban Sodium
- Group 2 (placebo) (Placebo Comparator): Placebo capsule (250mg) will be taken by mouth daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ifetroban Sodium — Given by mouth
  Arms: Group 1 (ifetroban)
Other: Placebo — Given by mouth
  Arms: Group 2 (placebo)

SUMMARY:
This pilot trial studies the side effects of ifetroban in treating patients with malignant solid tumors that are at high risk of coming back after treatment and spreading throughout the body. Platelets are a type of blood cells that help with clotting. Cancer cells stick to platelets and ride on them to get to different parts of the body. Drugs, such as ifetroban, may help these platelets become less "sticky," and reduce the chance of cancer cells spreading to other places in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of ifetroban sodium (ifetroban) administration in patients with malignant solid tumors at high risk of metastatic recurrence, after completion of all planned (neo)adjuvant locoregional and systemic therapies.

SECONDARY OBJECTIVES:

I. To assess rate of metastatic recurrence after completion of ifetroban in patients with malignant solid tumors.

EXPLORATORY OBJECTIVES:

I. To quantify pharmacodynamic markers of ifetroban effects.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 1 (IFETROBAN): Patients receive ifetroban sodium orally (PO) once daily (QD). Courses repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.

GROUP 2 (PLACEBO): Patients receive a placebo PO QD. Courses repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Subjects ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Current diagnosis of any stage I to III malignant solid tumor at high risk of metastatic recurrence (deemed by treating physician as patients with ≥ 50% chance of cancer metastatic recurrence within 5 years of diagnosis)
* Patients must have completed all standard locoregional and systemic therapy for their cancer within 120 days of study enrollment.
* Administration of an investigational agent prior to enrollment needs to be completed at least 30 days prior to enrollment
* Patients must have recovered (≤ grade 1 toxicities or grade 2 toxicities well managed with optimal medical care) from effects of local (surgery, radiation) or systemic treatments.
* Platelet count ≥ 100,000 per mL of blood
* Hemoglobin ≥ 9/g/dL (may have been transfused)
* Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min as calculated using the Cockcroft-Gault (CG) equation
* Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × ULN
* INR below upper limit of normal (ULN)
* Female patients of childbearing potential and non-sterile males must agree to use at least two methods of acceptable contraception from 15 days prior to first trial treatment administration until at least 5 months after study participant's final dose of study drug

Note: Females of childbearing potential are defined as those who are not surgically sterile or post-menopausal (i.e. patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrheic for 12 months without an alternative medical cause). Post-menopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone (FSH) level within laboratory reference range for postmenopausal women. Non-sterile males are those who have not had a vasectomy with documentation of the absence of sperm in the ejaculate.

* Patients unable to read/write in English are eligible to participate in the overall study but will not participate in the Patient-Reported Outcome questionnaires throughout the trial.
* Re-enrollment of a subject that has discontinued the study as a pre-treatment screen failure (i.e. a consented patient who did not receive study drugs) is permitted. If reenrolled, the subject must be re-consented. Only the screening procedures performed outside of protocol-specified timing must be repeated.

Exclusion Criteria:

* Evidence of biopsy-proven distant metastatic disease after completion of standard treatment
* Current use of anti-platelet drugs (ASA, NSAIDs, clopidogrel, argatroban, etc.) or anticoagulants (warfarin, heparin products, etc.)
* Active malignancy within 5 years prior to current diagnosis except for in situ disease or cancer with very high curability rate (i.e. testicular cancer, etc.)
* Uncontrolled co-morbid serious systemic illnesses that in the opinion of the investigator could compromise therapeutic safety.
* No concurrent anticancer therapy. Required washout from prior therapy:

  * Chemotherapy: 21 days
  * Major surgery: 14 days (provided wound healing is adequate)
  * Radiation: 7 days
  * Investigational/Biologic Therapy: 30 days
* Current symptomatic congestive heart failure (New York Heart Association > class II), unstable cardiac arrhythmia requiring therapy (e.g. medication or pacemaker), unstable angina (e.g. new, worsening or persistent chest discomfort), or uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100mmHg). Or any of the following occurring within 6 months (180 days) prior to first dose of study drugs: Myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack. (Use of antihypertensive medication to control blood pressure is allowed.)
* Ongoing peptic ulcer disease requiring treatment
* History of gastrointestinal bleed
* Severe gastro-esophageal reflux disease requiring treatment
* History of bleeding diathesis
* Pregnant or breastfeeding females.
* Prisoners or subjects who are involuntarily incarcerated.
* Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the patient's study physician to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with scheduled visits, treatment schedule, laboratory tests and other study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after completing treatment
Adherence to treatment (participants will be provided a pill diary to record when they take their medication. Study staff will collect the pill diary from participants at their clinic visits). | Up to 12 months
Summarized change of FACT-G score (scale = 0 to 4) | Up to 12 months

SECONDARY OUTCOMES:
Percentage of patients within metastatic recurrence (within each cohort) | At 12 months
Event-free survival (within each cohort) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Reid, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT03694249/ICF_000.pdf